CLINICAL TRIAL: NCT02111694
Title: Influence of Bottle-Type on Infant Feeding Behaviors
Acronym: OBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OBS-1303001967
Record Dates: First submitted 2014-03-26; First posted 2014-04-11 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Conventional Clear Bottle; Opaque Weighted Bottle
Keywords: infant; intake; satiation; mother; feeding practices; bottle feeding; formula feeding; maternal responsiveness; infant cues
MeSH Terms: conditions — Bottle Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Clear versus Opaque Bottle (Experimental): This is a within-subject study; all infants will be exposed to both conditions. Order of presentation will be counterbalanced across infants.
  Interventions: Behavioral: Bottle Type

INTERVENTIONS:
Behavioral: Bottle Type — Infants will be fed from a conventional, clear bottle during one feeding and from an opaque, weighted bottle from another feeding

SUMMARY:
The objective of the proposed research is to conduct a within-subject, experimental study that will describe mothers' feeding practices during typical bottle-feeding conditions and will examine whether removal of visual cues related to the amount of milk/formula in the bottle will alter these feeding practices. The investigators hypothesize that mothers will show higher levels of infant-directed feeding practices and lower levels of mother-directed feeding practices when using opaque, weighted bottles compared to when using standard, clear bottles. The investigators also hypothesize that infants will consume less breast milk or formula when fed from opaque, weighted bottles compared to when fed from standard, clear bottles.

ELIGIBILITY:
Inclusion Criteria:

* Mothers must be 18 years or older
* Infants must be between 0- and 6-months of age
* Infants must be prior to the introduction of solid foods

Exclusion Criteria:

* Preterm birth
* Medical conditions that interfere with feeding

Max Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2013-06; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Infant intake within a feeding (mL) | 3-hour period
  assessed by weighing the bottle before and after a feeding
Maternal responsiveness to infant cues during a feeding | 3-hour period
  assessed by the Nursing Child Assessment Satellite Training Parent-Child Interaction Feeding Scale

SECONDARY OUTCOMES:
Maternal perception/acceptance of the bottles during a feeding | 3-hour period

CONTACTS AND LOCATIONS:
Overall Officials: Alison K Ventura, PhD, Principal Investigator — Drexel University
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Ventura AK, Pollack Golen R. A pilot study comparing opaque, weighted bottles with conventional, clear bottles for infant feeding. Appetite. 2015 Feb;85:178-84. doi: 10.1016/j.appet.2014.11.028. Epub 2014 Nov 28. PMID 25445988
- [Derived] Golen RB, Ventura AK. Mindless feeding: Is maternal distraction during bottle-feeding associated with overfeeding? Appetite. 2015 Aug;91:385-92. doi: 10.1016/j.appet.2015.04.078. Epub 2015 May 4. PMID 25953601